CLINICAL TRIAL: NCT03870321
Title: Efficacy of Core Training to Improve Abdominal Strength Strength and Analyze Whether it Provides Improvement in Ankle Proprioception in Federated Basketball Players From 18 to 40 Years: A Pilot Study
Brief Title: Core Training to Improve Abdominal Strength Strength and Ankle Proprioception in Basketball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Strength
Record Dates: First submitted 2019-03-08; First posted 2019-03-12 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Proprioceptive Disorders
Keywords: Core; Strength; Proprioception; Ankle; Basketball
MeSH Terms: conditions — Somatosensory Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core training (Experimental): The subjects who are in the experimental group will carry out the Core training routine
  Interventions: Other: Core training
- Control (No Intervention): The subjects who are in the control group will not receive intervention and will continue with their daily routine and training

INTERVENTIONS:
Other: Core training — In the first week different types of abdominal exercises will be performed: standard, with trunk rotation, extension of the back raising the upper extremity of the body and legs, extension of the back raising one arm and the contralateral leg. In the same way, the subject will raise from the quadruped position one arm and the contralateral leg on each side, and we will ask for the exercise of the front plate, positioning itself in a position of four support points: feet and elbows. When performing the rear bridge exercise the subject will raise the trunk resting on both feet, while in the lateral bridge exercise will be done with support on the right and left side. All exercises will be done for 30 seconds, in 3 series).
  During the next three weeks we will continue with the same training, but for each week we will increase 10 seconds per exercise.
  Arms: Core training

SUMMARY:
Introduction. The prevalence of ankle injuries in basketball are high. The lack of balance in the ankle is one of the main causes that produces these injuries. The goal of core training is to increase the physical capacities of resistance strength in the abdomen and analyze if it produces improvement in proprioception in the ankle joint in basketball players.

Objective. To evaluate the effectiveness of Core training to improve the strength of the abdomen and analyze if it produces improvement in proprioception in ankle of basketball players.

Study design. Randomized, multicentric, single-blind clinical study with a follow-up period.

Methods. The 30 participants recruited will be randomly assigned to the two study groups: experimental (Core training for strength in the abdomen) and control (without intervention). The treatment will last 4 weeks, with 3 weekly sessions, approximately 20 minutes each. There will be three evaluations (pre-intervention, post-intervention and follow-up). On the dependent variables: strength core resistance (evaluated with Trunk Flexor Test, Trunk Extender Test, and Side Bridge Test) and proprioception (measured with the Star Excursion Balance tests and Romberg test) With the Kolmogorov Smirnov statistical test we will calculate the normality and with the t-student test of paired data and an ANOVA of repeated measures, we will obtain the difference between the three evaluations and the intra and intersubject effect, respectively.

Expected results. To observe improvement in strength in the abdomen and analyze if it produces improvement in proprioception in the ankle of basketball players.

ELIGIBILITY:
Inclusion Criteria:

* Basketball players
* Federated in the Community of Madrid
* Male
* With an age range of 18 to 40 years.

Exclusion Criteria:

* Who have a musculoskeletal injury at the time of the study or who have suffered a lower limb injury in a period of three months before the study
* That they are in an individualized personal training
* Not signed the informed consent document.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline ankle proprioception after intervention and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The Star excursion balance test will be used to measure ankle proprioception. It begins with a star drawn on the ground, while the subject will remain in a static position, placing his or her bare foot in the center of the star. During the execution of the test the subject will be asked to touch the farthest point possible with the tip of the first finger. The contact of the finger has to be clean, without supporting the weight or imbalance of the other foot, returning each time to the initial monopodal position. At each attempt the contact point will be recorded on the ground line. This exercise will be repeated three times and the average of the evaluations will be taken into account to obtain the value of the measurement in each one of the directions to be studied, with the final result being the average distance of all the attempts in each of the directions. The unit of measurement is the centimeter (the greater distance in centimeters, the better ankle proprioception).

SECONDARY OUTCOMES:
Change from baseline strength of the flexor muscles of the abdomen after intervention and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The Trunk Flexor Test will be used to measure the strength of the flexor muscles of the abdomen. The subject will be sitting on a bench, with knees and hips bent at 90 degrees and feet tied to the stretcher. The arms should be crossed over the chest and trunk in a flared position at 60 degrees. The subject must maintain that position as long as possible. The test is terminated when the participant can not sustain the initial position. The unit of measure is temporary (seconds). The greater the amount of time, the greater the strength of the flexor muscles of the abdomen.
Change from baseline strength of the extensor muscles of the abdomen after intervention and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  Researchers will use the Trunk Extender Test to evaluate the strength of the extensor muscles of the abdomen. The athlete will be placed in prone position, with the pelvis and ankles fixed to the stretcher with a strap, with the navel on the edge of the stretcher. A chair should be placed at the same height as the stretcher to support the trunk and upper extremity. Then the chair will be removed and the subject should maintain a horizontal position with arms crossed to the trunk as long as possible. The test ends when the subject can not hold the initial position anymore and touch the chair in front of them with their hands. The unit of measure is temporary (seconds). The greater the amount of time, the greater the strength of the extensor muscles of the abdomen.
Change from baseline strength of the lateral flexor muscles of the abdomen after intervention and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The Side Bridge Test will be used to measure the strength of the lateral flexor muscles of the abdomen. The subject will be placed in the lateral decubitus with the knees extended on the stretcher being asked to lift the hip of the stretcher using only the feet and the elbow as support. The test will end when the hip falls. The unit of measure is temporary (seconds). The greater the amount of time, the greater the strength of the lateral flexor muscles of the abdomen.
Change from baseline ankle proprioception after intervention and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The Romberg test will be used to measure proprioception. The athlete will be asked to stand with their feet together, their arms loose on their sides and their eyes open. In this position any imbalance will be recorded and subsequently you will be asked to close your eyes. The stability will be observed and it will be compared with the one presented with the eyes open. The degree of oscillation and the direction of hips, knees and the entire body should be evaluated. The test is considered positive if there is an imbalance or if the oscillation worsens significantly with the closing of the eyes (score 1). Otherwise, it will be negative (score 0).

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Universidad Europea de Madrid, Madrid, Comunity of Madrid, Spain